CLINICAL TRIAL: NCT07286760
Title: Comparison of the Effects of MAT Pilates and MIHA Combined Exercise Programs on Pain, Quality of Life, Anxiety, and Endurance in Patients With Nonspecific Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-78097791-020-4745
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
Keywords: exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIHA Combined Exercise Programs (Experimental)
  Interventions: Other: MIHA Combined Exercise Programs
- MAT Pilates (Active Comparator)
  Interventions: Other: MAT Pilates

INTERVENTIONS:
Other: MIHA Combined Exercise Programs — MIHA Combined Exercise Programs
  Arms: MIHA Combined Exercise Programs
Other: MAT Pilates — MAT Pilates
  Arms: MAT Pilates

SUMMARY:
Comparison of the Effects of MAT Pilates and MIHA Combined Exercise Programs on Pain, Quality of Life, Anxiety, and Endurance in Patients with Nonspecific Back Pain

ELIGIBILITY:
Inclusion Criteria:

Being between 25 and 45 years of age Having had back pain for the last 3 months The back pain not being due to a structural, traumatic, infectious, or tumor-related cause (i.e., no specific cause has been identified) Not having any serious cardiovascular, neurological, or orthopedic conditions that would prevent participation in a physical exercise program Not having participated in a regular physical exercise program in the past 6 months Not having any contraindications to the use of a wearable EMS device (e.g., not having a pacemaker)

Exclusion Criteria:

The back pain is associated with a specific pathology (e.g., spinal stenosis, fracture, tumor, infection, etc.) Being within the first 6 months of pregnancy or postpartum History of neurological disease (e.g., multiple sclerosis, peripheral neuropathy, spinal cord injury, etc.) Having a pacemaker or other electronic device in the body Pre-existing intolerance to EMS

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | 12 weeks
  An algometer will be used to measure pain levels. We have identified three muscle groups for the algometer: Gluteus Medius, Erector Spinae, and Quadratus Lumborum. A low level indicates greater sensitivity and weakness.
Quality of Life Assessment | 12 weeks
  Quality of life will be assessed using the Oswestry Disability Index. It is used to evaluate the effect of the MAT Pilates and EMS-assisted exercise programs applied in the study on daily living activities. The lower the total score, the less the disability.
Anxiety Assessment | 12 weeks
  Individuals' anxiety levels are assessed using the Beck Anxiety Scale. This assessment aims to compare individuals' anxiety levels before and after intervention. A high score on the Beck Anxiety Scale indicates a higher level of anxiety.
Endurance Assessment | 12 weeks
  : Individual endurance is assessed using three movements: the Plank, Bridge Movement, and V-Sit position. These selected movements target the anterior, posterior, and lateral core muscle groups, enabling an assessment of overall endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazal GENÇ, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No